CLINICAL TRIAL: NCT01759121
Title: Randomized, Parallel Controlled, Clinical-trial on 532nm Laser Partially Subthreshold Panretinal Photocoagulation With PASCAL Endpoint Management Function for Severe Non-proliferative Diabetic Retinopathy(NPDR)
Brief Title: Safety and Effectiveness Study of 532nm Laser Subthreshold Panretinal Photocoagulation for Severe NPDR
Acronym: S-PRP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jin Chen-jin, Dr, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S-PASCAL-PRP; ChiCTR-TRC-12002735 (Registry Identifier: Chinese Clinical Trial Registry)
Record Dates: First submitted 2012-12-18; First posted 2013-01-02 (Estimated); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: Severe Non-proliferative Diabetic Retinopathy
Keywords: severe non-proliferative diabetic retinopathy; subthreshold; panretinal photocoagulation; PASCAL; endpoint management

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- T-PRP (Active Comparator): 532nm-short pulse panretinal photocoagulation with PASCAL function
  Interventions: Radiation: T-PRP
- S-PRP (Experimental): 532nm-partially subthreshold short pulse panretinal photocoagulation with PASCAL endpoint management function
  Interventions: Radiation: S-PRP

INTERVENTIONS:
Radiation: T-PRP — 532nm-short pulse panretinal photocoagulation with PASCAL function
  Other Names: Traditional-PRP
  Arms: T-PRP
Radiation: S-PRP — 532nm-partially subthreshold short pulse panretinal photocoagulation with PASCAL endpoint management function
  Other Names: Subthreshold PRP
  Arms: S-PRP

SUMMARY:
This randomized, parallel controlled, clinical-trial aims to evaluate the therapeutic efficacy of 532nm laser partially subthreshold panretinal photocoagulation with PASCAL endpoint management function for severe non-proliferative diabetic retinopathy.

DETAILED DESCRIPTION:
This randomized, parallel controlled, clinical-trial aims to evaluate the therapeutic efficacy of 532nm laser partially subthreshold panretinal photocoagulation with PASCAL endpoint management function for severe non-proliferative diabetic retinopathy : (1)To evaluate therapeutic effect of 532nm laser partially subthreshold panretinal photocoagulation with PASCAL endpoint management function for severe non-proliferative diabetic retinopathy; (2)To compare side effect of 532nm laser partially subthreshold panretinal photocoagulation with PASCAL endpoint management function on retina with traditional visible endpoint panretinal photocoagulation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of severe non-proliferative diabetic retinopathy
* Age:45-80 years
* Best corrected visual acuity(BCVA) ≥20/100,Myopia≤-6 degree(-6D)
* No photocoagulation (PRP) before this clinical trial and no major ocular surgery (including cataract extraction, or any other intraocular surgery) within 3 months
* Ability and willingness to provide informed consent

Exclusion Criteria:

* Participate in other clinical trials within 3 months
* Severe refractive media turbidity; Unable to accept laser treatment such as nystagmus, etc
* Medically or mentally unstable(including cardiovascular disorders, cerebrovascular diseases,liver and kidney disease,hematological disorder and psychosis
* Conditions that in the opinion of the investigator would interfere trial results or increase risk
* Conditions that in the opinion of the investigator would preclude participation in the study

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2016-03 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
change of best corrected visual acuity | 1 year
  best corrected visual acuity
the probability of vitreous haemorrhage | 1 year

SECONDARY OUTCOMES:
Central Retinal Thickness | 1 year
foveal volume of macula | 1 year
amount of microaneurysms | 1 year
amount of bard exudate | 1 year
amount of retinal hemorrhage | 1 year
amount and area of IRMA | 1 year
amount of neovascularization | 1 year
change of ischemia area | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Chen-jin Jin, Study Director — Zhongshan Ophthalmic Center, Sun Yat-sen University; Pei-pei Wu, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Li Z, Lu T, Zhou L, Huang C, Zhao H, Liang J, Li C, Cong Q, Lan Y, Jin C. Retinal and Choroidal Alterations in Diabetic Retinopathy Treatment using Subthreshold Panretinal Photocoagulation with Endpoint Management Algorithm: A Secondary Analysis of a Randomized Clinical Trial. Ophthalmol Ther. 2023 Aug;12(4):1867-1880. doi: 10.1007/s40123-023-00713-0. Epub 2023 Apr 30. PMID 37120774
- [Derived] Zhao H, Zhou L, Lai K, Yu M, Huang C, Xu F, Li C, Lu L, Jin C. Comparison of functional changes of retina after subthreshold and threshold pan-retinal photocoagulation in severe non-proliferative diabetic retinopathy. Lasers Med Sci. 2022 Dec;37(9):3561-3569. doi: 10.1007/s10103-022-03635-8. Epub 2022 Sep 7. PMID 36070046
- See also: a clinical study on subthreshold panretinal photocoagulation for proliferative diabetic retinopathy (PDR) — http://www.nature.com/eye/journal/v22/n5/full/6702725a.html